CLINICAL TRIAL: NCT06058962
Title: A Three-Arm, Prospective, Randomized, Double Blind, Placebo-Controlled Trial Evaluating the Efficacy and Safety of 2 Doses of Suramin vs. Placebo in Male Children With ASD Receiving Standard Treatment
Brief Title: Double Blind Trial in Children With Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paxmedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUR-ONQ-ASD-001
Record Dates: First submitted 2023-09-18; First posted 2023-09-28 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Suramin

STUDY DESIGN:
Intervention Model Description: The participants were randomized to one of three double-blind treatment groups, i.e., Arm A (10 mg/kg suramin) or Arm B (20 mg/kg suramin) or Arm C (placebo) in a targeted 1:1:1 ratio, as per the randomization schedule and stratification plan. The stratification plan was to match patients by age (< 7 vs ≥ 7), ADOS-2 comparison scores (≤ 8.5 vs > 8.5) and NVIQ (≤ 80 vs > 80)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was double-blind. Suramin and placebo are both clear solutions when prepared.
  Suramin was prepared by an unblinded pharmacist by reconstituting 1 g vial of suramin in 10 mL of sterile water for infusion to prepare a 10% (100 mg/mL) solution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suramin 10 mg/kg (Experimental): 50 mg test dose of suramin (upon first administration), then suramin 10 mg/kg (minus 50 mg suramin test dose) in 50 mL of saline administered by IV infusion over 30 minutes was given at Visits 2, 4, and 5.
  Interventions: Drug: Suramin Sodium
- Suramin 20 mg/kg (Experimental): 50 mg test dose of suramin (upon first administration), then suramin 20 mg/kg (minus 50 mg suramin test dose) in 50 mL of saline administered by IV infusion over 30 minutes was given at Visits 2, 4, and 5.
  Interventions: Drug: Suramin Sodium
- Placebo (Placebo Comparator): Test dose of saline placebo, then saline placebo infusion of 50 mL administered over 30 minutes was given at Visits 2, 4, and 5.
  Interventions: Drug: Suramin Sodium

INTERVENTIONS:
Drug: Suramin Sodium — Suramin sodium is a sodium salt form of suramin, an antitrypanosomal compound.
  Other Names: Placebo

SUMMARY:
This study investigated the safe and efficacious use of suramin as a novel treatment for ASD by testing two suramin doses vs placebo

DETAILED DESCRIPTION:
PUR-ONQ-ASD-001 was a multicenter, 3-arm, prospective, randomized, double blind, placebo-controlled multiple dose trial involving 2 dose levels of suramin vs. placebo. The study randomized 52 male participants who received treatment interventions for ASD; each treatment arm was assigned approximately 17 participants. The number of participants was increased to 52 participants (48 originally planned) due to early withdrawals related to the COVID-19 global pandemic lockdowns and other matters. Participants were stratified by age, ADOS-2, and Non-verbal Intelligence Quotient (NVIQ). Participants who met all the inclusion criteria and none of the exclusion criteria were randomized through an electronic system to either arm A (10 mg/kg suramin) or Arm B (20 mg/kg suramin) or Arm C (Placebo) in a targeted 1:1:1 ratio, as per the randomization schedule and stratified by age, ADOS-2, and NVIQ. All participants received a 50 mg test dose at their first administration (0.5 mL of freshly reconstituted 10% solution in 5 mL saline) to check for allergic reactions. The test dose was given by slow intravenous (IV) infusion for 30 minutes then flushed with 10 mL saline. Vitals were checked for 30 min and if there were no changes or evidence of allergic reaction, the rest of the study drug dose was administered (10 mg/kg or 20 mg/kg minus test dose [minus 50 mg] in a 50 mL saline up to a maximum of 1 g given over 30 minutes). Arm A - 50 mg test dose of suramin (upon first administration), then suramin 10 mg/kg (minus 50 mg suramin test dose) in 50 mL of saline administered by IV infusion over 30 minutes was given at Visits 2, 4 and 5. The maximum dose administered was 1 g.

Arm B - 50 mg test dose of suramin (upon first administration), then suramin 20 mg/kg (minus 50 mg suramin test dose) in 50 mL of saline administered by IV infusion over 30 minutes was given at Visits 2, 4 and 5. The maximum dose administered was 1 g.

Arm C - Test dose of saline placebo, then saline placebo IV infusion of 50 mL administered over 30 minutes was given at Visits 2, 4 and 5

ELIGIBILITY:
Inclusion Criteria:

* Male children aged 4 - 17 years
* Participants with or without treatment interventions for ASD
* Participants must have been diagnosed with ASD by Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V)
* Autism diagnostic observation schedule, version 2 (ADOS-2) Comparison scores in the
* moderate and high level as evaluated on the ADOS-2
* Stable treatment intervention for ≥ 2 months
* Participants agreed to not change their treatment interventions throughout the study
* duration
* Participants on Ritalin and Risperdal or similar medication agreed to not change their
* dose during the study

Exclusion Criteria:

* Hospitalization within the previous 2 months
* An acute medical problem, Rett syndrome, microcephaly, tuberous sclerosis, neurofibromatosis, epilepsy, or clinically significant liver, kidney, or adrenal disease or persons suffering from any serious acute condition where, in the investigator's opinion, the participant's well-being may have been compromised
* Planning to start a new drug, diet, or behavioral intervention during the study
* Weight under the 5th percentile for age
* Unable to tolerate venipuncture, urine collection, or an indwelling IV catheter for 3-4 hours
* Plasma creatinine above normal for age and weight according to the laboratory reference ranges.
* Liver function alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5-fold above the upper limit of normal
* Known intolerance to suramin or other antipurinergic drugs
* Unable to perform or cooperate with study requirements
* Children with known syndromic forms of ASD caused by DNA mutation or chromosomal copy number variation

Ages: 4 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Males only
Enrollment: 52 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
The primary objective was to evaluate the safety of 2 dose levels of low-dose suramin against placebo in children with ASD receiving standard treatment. | 98 Days
  Adverse Events and Laboratory Results

SECONDARY OUTCOMES:
The primary objective was to evaluate the efficacy of 2 dose levels of low-dose suramin against placebo in children with ASD receiving standard treatment. | 98 Days
  Aberrant Behavior Checklist (ABC) and (Clinical Global Impression) CGI scales used to evaluate efficacy.
  ABC scoring is a 0 as improvement with a 3 as a problem being severe.
  For each item, decide whether the behavior is a problem for your child/adolescent and select the appropriate number/response:
  "0 = not at all a problem
  1. = the behavior is a problem but slight in degree
  2. = the problem is moderately serious
  3. = the problem is severe in degree

CONTACTS AND LOCATIONS:
Overall Officials: jennifer L bonfrisco, Study Director — Paxmedica
Locations (1):
- PaxMedica, Tarrytown, New York, United States

IPD SHARING:
Plan to Share IPD: No
Abstract and CSR

REFERENCES:
- [Derived] Hough D, Mao AR, Aman M, Lozano R, Smith-Hicks C, Martinez-Cerdeno V, Derby M, Rome Z, Malan N, Findling RL. Randomized clinical trial of low dose suramin intravenous infusions for treatment of autism spectrum disorder. Ann Gen Psychiatry. 2023 Nov 6;22(1):45. doi: 10.1186/s12991-023-00477-8. PMID 37932739